CLINICAL TRIAL: NCT00131651
Title: A Dose-Ranging, Phase II, Open Label Study of ATN 161 in Advanced Renal Cell Cancer
Brief Title: ATN-161 in Advanced Renal Cell Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Attenuon (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATN-161-005
Record Dates: First submitted 2005-08-17; First posted 2005-08-19 (Estimated); Last update posted 2007-12-06 (Estimated); Status verified 2007-12

CONDITIONS: Carcinoma, Renal Cell
Keywords: renal; cancer; advanced; unresectable; metastatic; recurrent; anti-angiogenic; targeted; ATN-161; Recurrent renal cell cancer; Renal clear cell carcinoma; Advanced Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms; Neoplasm Metastasis; Recurrence | interventions — acetyl-prolyl-histidyl-seryl-cysteinyl-asparaginamide

INTERVENTIONS:
Drug: ATN-161

SUMMARY:
The purpose of this study is to determine an active dose of ATN-161 for future studies while establishing preliminary evidence of effectiveness in patients with renal cell cancer.

DETAILED DESCRIPTION:
Angiogenesis, defined as the growth of new blood vessels from pre-existing vessels, is a requirement for the growth of nearly all tumors. Clear cell renal cell carcinoma (CCRCC) is a malignancy characterized by abundant vascularization and a high degree of resistance to chemotherapy which makes antiangiogenic therapy an intriguing concept for treatment. This concept has been established by the initial successes observed in recent studies of antiangiogenic therapies for CCRCC. ATN-161 is an attractive candidate for investigation as a therapeutic agent in CCRCC because it binds to several fully activated integrins, which are essential downstream components in the angiogenic signaling cascade.

Functional imaging using dceMRI has been demonstrated as an effective way to show effects on the vasculature across different tumors, including CCRCC. Preclinical experiments have shown that ATN-161 affects tumor perfusion in tumor bearing mice. Therefore, use of imaging in this study is expected to be an effective method for evaluating the antiangiogenic response to ATN-161.

Patients will be administered ATN-161 three times weekly by short (10 minute) IV infusion at 1 of 3 dose levels (20, 100, and 600 mg). Patients will be treated until progression of disease, unacceptable drug toxicity, or withdrawal of consent occurs.

Functional imaging (dceMRI) will be performed within 1 week prior to first treatment, again during the second week of treatment, and finally during the fourth week of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have unresectable and/or metastatic kidney cancer with a component of clear cell adenocarcinoma that is histologically confirmed. A pathologist at the investigator's institution must have reviewed the material sent by outside institutions and confirm the diagnosis.
2. Patients must have been previously treated with at least one FDA-approved therapy or commonly used treatment (such as interferon or low dose interleukin-2) for advanced kidney cancer. Any number of other prior treatments, approved or investigational, is acceptable.
3. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as 2 times the measurable slice width with spiral CT scan. See RECIST Appendix B for the evaluation of measurable disease.
4. Patients must have at least one lesion amenable to dceMRI as per lesion guidelines (see Section 8.1.1).
5. Age ≥18 years.
6. ECOG performance status of 0 or 1 (see Appendix A).
7. Patients must have recovered from the reversible effects of prior treatment (with the exception of alopecia) by returning to normal or mild severity (Grade 1) or their pre-treatment baseline.
8. Life expectancy of greater than three months.
9. Patients must have adequate organ and marrow function as defined below:

   * absolute neutrophil count ≥1,500 cells/mm3
   * platelets ≥100,000 cells/mm3
   * total bilirubin ≤1.5 mg/dL
   * AST (SGOT) and ALT (SGPT) ≤1.5 x institutional upper limit of normal (ULN) (≤2.5 x ULN for patients with liver metastases)
   * alkaline phosphatase ≤5.0 x ULN
   * serum creatinine ≤1.5 x ULN
   * serum calcium ≤1 x ULN (the patient may be on treatment for hypercalcemia)
10. The effects of ATN 161 on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because antiangiogenic agents are known to be teratogenic, women of child-bearing potential and men with partners of child-bearing potential must agree to use adequate contraception (hormonal and/or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation through the follow up visit 28 days after the last dose of ATN 161. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Similarly, if the partner of a male patient should become pregnant while he is participating in this study, he should inform his treating physician immediately.
11. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who have not recovered from reversible adverse events due to previously-administered agents.
2. Patients may not be receiving any agents, approved or investigational, for the treatment of CCRCC, and may not be receiving any investigational agents for other conditions.
3. Patients with documented brain metastases are excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Institutional practices should be followed to establish the absence of brain metastases.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
5. Pregnant women are excluded from this study because ATN 161 is an antiangiogenic agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ATN 161, breastfeeding should be discontinued if the mother is treated with ATN 161.
6. Patients known to be human immunodeficiency virus (HIV)-positive are excluded.
7. Patients who cannot undergo dceMRI analysis for any reason.
8. Patients who do not have adequate wound healing based on clinical judgment following a major surgical intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2005-08

PRIMARY OUTCOMES:
Reduction in tumor blood flow and permeability of vessels

SECONDARY OUTCOMES:
Response rate (time to progression, rate of objective response, and rate and duration of disease control)
Safety (adverse events [AEs], lab tests and physical examinations)
Reduction in circulating endothelial cells (CECs)
Reduction in circulating endothelial progenitor cells (CEPs)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of California Irvine, Chao Family Comprehensive Cancer Center, Irvine, California
  - University of California San Francisco Comprehensive Cancer Center, San Francisco, California
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin